CLINICAL TRIAL: NCT07308587
Title: Prospective Evaluation of Intercostal Neuralgia Incidence, Risk Factors, and Outcomes in Patients With Chest Tube Insertion After Traumatic Rib Fractures
Brief Title: Evaluation of Intercostal Neuralgia in Patients With Chest Tube Insertion After Traumatic Rib Fracture
Status: Not yet recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: SUN 6775
Record Dates: First submitted 2025-09-05; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-09

CONDITIONS: Intercostal Nerve Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chest tube inserted: Patients with acute traumatic rib fracture/chest injury requiring chest tube insertion
  Interventions: Procedure: Chest tube insertion

INTERVENTIONS:
Procedure: Chest tube insertion — Insertion of chest tube

SUMMARY:
Traumatic rib fractures are common injuries following blunt chest trauma, often requiring chest tube insertion to manage complications such as pneumothorax or haemothorax. However, chest tube placement can lead to intercostal nerve injury, resulting in intercostal neuralgia-a debilitating condition characterized by chronic, neuropathic pain along the intercostal nerves. Despite its clinical significance, the incidence, risk factors, and long-term outcomes of intercostal neuralgia in this patient population remain poorly understood.

Chronic pain following thoracic trauma, including intercostal neuralgia, has been shown to significantly impair quality of life and functional outcomes, leading to prolonged disability and increased healthcare utilization. Current literature highlights the need for better understanding and management of this condition, particularly in patients undergoing invasive procedures such as chest tube insertion. This study aims to prospectively evaluate the development of intercostal neuralgia in patients with chest tube insertion following traumatic rib fractures.

DETAILED DESCRIPTION:
Intercostal neuralgia is defined as pain along the intercostal nerve distribution with neuropathic features. Chronic intercostal neuralgia is defined as having intercostal neuralgia symptoms for >3 months.

Intercostal neuralgia pain will be specifically differentiated from persistent rib fracture pain through the presence of neuropathic pain at the level of the chest tube/pigtail that is reproducible with brushing/light touch to the chest tube scar site.

The following data will be collected:

Baseline:

* Demographic information (age, sex, ethnicity, comorbidities).
* Pain assessment using numerical rating scale at rest and with deep inspiration
* Pre-existing chronic pain conditions (e.g., fibromyalgia, chronic regional pain syndrome) and history of prior thoracic surgery or chest tube insertion.
* Injury characteristics (mechanism of injury including presence of foreign bodies and additional penetrating injuries, number and location of rib fractures, associated injuries including vertebral body fractures, sternal fracture, transverse process fracture).
* Chest tube / pigtail details (size, insertion site, duration of placement).
* Spirometry testing including forced vital capacity (FVC) and forced expiratory volume (FEV1) at time of enrolment of study

Additional information to be collected following hospital stay:

* Analgesic use including dose of opioids, use of regional anesthesia techniques, and adjunct analgesic medications while in hospital
* Length of hospital stay
* Presence and duration of mechanical ventilation
* Number of surgeries

Follow ups: 1 (± 3 days) and 3 months (± 1 week) via telephone

* Pain assessment using the numerical rating scale at rest and with deep inspiration
* S-LANSS for neuropathic pain
* EQ-5D-5L for health related quality of life
* PROMIS sleep disturbance 6a for sleep
* Medication use (analgesics, neuropathic pain medications)

Patients who are found to have intercostal neuralgia at 3 month follow up assessment can be referred to the pain clinic and choose to be sent for formal ultrasound to identify and characterize findings to indicate the presence of neuroma (a non-cancerous tumor or growth of nerve tissue), degree of scarring, or any other pain generating causes, if agreed. Participants' preferences regarding the disclosure of neuroma, including their right to know or not to know, will be respected (as described in the consent form).

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with traumatic rib fractures requiring chest tube insertion
* Chest tube or pigtail insertion performed during their initial hospitalization for trauma

Exclusion Criteria:

* Patients with traumatic brain injury
* Patients with spinal cord injury
* Inability to complete follow-up assessments (e.g., language barriers, lack of telephone access)

Exclusion Criteria:

* Patients with traumatic brain injury
* Patients with spinal cord injury
* Inability to complete follow-up assessments (e.g., language barriers, lack of telephone access)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute traumatic rib fractures requiring chest tube insertion for management.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of intercostal neuralgia | 1 and 3 months
  To determine the incidence of intercostal neuralgia in patients undergoing chest tube insertion after traumatic rib fractures. Presence of neuropathic pain to be assessed using S-LANSS

SECONDARY OUTCOMES:
Assess the impact of intercostal neuralgia on quality of life and functional outcomes | 1 and 3 months
  Assess the impact of intercostal neuralgia on quality of life using EQ-5D-5L
Assess the impact of intercostal neuralgia on quality of life and functional outcomes | 1 and 3 months
  Assess the impact of intercostal neuralgia on quality of life using Promis 6a Sleep questionnaire
Assess the impact of intercostal neuralgia on medication use | 1 and 3 months
  Determine the impact of intercostal neuralgia on medication use including opioids and anti-neuropathic medications by collection and assessment of quantity of medications taken for pain relief related to intercostal neuralgia.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bulger EM, Arneson MA, Mock CN, Jurkovich GJ. Rib fractures in the elderly. J Trauma. 2000 Jun;48(6):1040-6; discussion 1046-7. doi: 10.1097/00005373-200006000-00007. PMID 10866248
- [Result] Karmakar MK, Ho AM. Acute pain management of patients with multiple fractured ribs. J Trauma. 2003 Mar;54(3):615-25. doi: 10.1097/01.TA.0000053197.40145.62. PMID 12634549
- [Result] Bailey RC. Complications of tube thoracostomy in trauma. J Accid Emerg Med. 2000 Mar;17(2):111-4. doi: 10.1136/emj.17.2.111. PMID 10718232
- [Result] Fabricant L, Ham B, Mullins R, Mayberry J. Prolonged pain and disability are common after rib fractures. Am J Surg. 2013 May;205(5):511-5; discusssion 515-6. doi: 10.1016/j.amjsurg.2012.12.007. PMID 23592156
- [Result] Blyth FM, March LM, Brnabic AJ, Cousins MJ. Chronic pain and frequent use of health care. Pain. 2004 Sep;111(1-2):51-8. doi: 10.1016/j.pain.2004.05.020. PMID 15327808